CLINICAL TRIAL: NCT02890420
Title: Nutritional Status Of Under-Six Children: Epidemiology Study (NUTRI-STAT)
Acronym: NUTRI-STAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-01Obs-CHRMT
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Children Behavior About Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female children: Female children in third year of preschool in Thionville (north-eastern France)
- Male children: Male children in third year of preschool in Thionville (north-eastern France)

SUMMARY:
This study permit to evaluate the characteristics of children in third year of preschool, during a year, in 16 schools in Thionville (north-eastern France) by the way of the annual medical visit.The aim of the study is to describe the nutritional status of children under-six years of age: underweight, overweight, and obesity considering the sex. .

DETAILED DESCRIPTION:
For several decades the eating behavior has been changing. That note is obviously more true for children, with the arrival of new recipes, not really healthier for all. This study permit to evaluate the characteristics of children in third year of preschool, during a year, in 16 schools in Thionville (north-eastern France) by the way of the annual medical visit. The aim of the research is to estimate the healthy weight corresponding with a height considering the gender.

ELIGIBILITY:
Inclusion Criteria:

* third year of preschool in Thionville
* information of the legal responsibles

Exclusion Criteria:

* opposition of the legal responsible for gathering data

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in third year of preschool in one of the 16 schools in Thionville, Lorraine, FRANCE
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Body mass index of children | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CUNY, MD, Principal Investigator — CHR Metz-Thionville

IPD SHARING:
Plan to Share IPD: No